CLINICAL TRIAL: NCT07305779
Title: A Phase 1, Open-label, Single-sequence Pharmacokinetic Trial to Assess the Effect of a Single Oral Dose of SEP-380135 on the Potential for Cytochrome P4502D6 Mediated Drug-drug Interactions in Healthy Adults
Brief Title: A Trial to Test the Effects of Other Drugs on SEP-380135 in Healthy Men and Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 384-201-00004
Record Dates: First submitted 2025-12-12; First posted 2025-12-26 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-11

CONDITIONS: Schizophrenia
Keywords: Mental Health Conditions; Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — quinidine gluconate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SEP-380135 + Quinidine Gluconate (Experimental): Participants receive SEP-380135 alone on Day 1, followed by administration of quinidine gluconate beginning on Day 6. On Day 7, SEP-380135 is coadministered with quinidine gluconate. Quinidine gluconate dosing continues from Day 8 to Day 10.
  Interventions: Drug: SEP-380135; Drug: Quinidine Gluconate

INTERVENTIONS:
Drug: SEP-380135 — Oral capsules.
Drug: Quinidine Gluconate — Oral extended-release (ER) tablets.

SUMMARY:
The purpose of this study is to assess the effect of cytochrome P450 isoenzyme 2D6 (CYP2D6) inhibition by quinidine on the pharmacokinetic (PK) parameters of a single dose SEP-380135 in healthy adult participants.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants between 18 and 55 years of age (inclusive) at time of consent
2. Body mass index from 18.0 to 32.0 kilograms per square meter (kg/m^2) (inclusive).
3. In good health as determined by:

   1. Medical history
   2. Physical examination
   3. Vital signs
   4. Neurological examination
   5. Electrocardiogram
   6. Serum chemistry, lipid panel, thyroid panel, coagulation panel, urinalysis, hematology, and serology tests (from screening visit).
4. Willing to stay in the clinic for the required period (i.e., to be hospitalized for 10 days) and willing to be contacted for the safety follow-up telephone call.
5. Ability to provide written, informed consent prior to initiation of any trial-related procedures, and ability, in the opinion of the Principal Investigator, to comply with all the requirements of the trial.

Exclusion Criteria:

1. Have taken an investigational drug within 30 days or 5 half-lives, if known, (whichever is longer) prior to screening.
2. Have had previous exposure to SEP-380135.
3. Are currently participating in another clinical trial.
4. Attempted suicide within 12 months prior to screening.
5. A history of sick sinus syndrome, first-, second-, or third-degree atrioventricular block, myocardial infarction, New York Heart Association Class II-IV heart failure, cardiomyopathy, pulmonary congestion, cardiac arrhythmia, prolonged QT interval, congenital long QT syndrome, family history of long QT, or moderate to severe hypokalemia. A participant with non-clinically significant ECG abnormalities at screening and check-in requires approval from the medical monitor and the sponsor's physician.
6. In the opinion of the investigator, should not participate in the trial.

Note: Other protocol-specified inclusion/exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2025-03-07 (Actual); Primary Completion 2025-05-03 (Actual); Study Completion 2025-05-03 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Concentration (Cmax) of SEP-380135 and its Metabolites | Up to Day 11
Area Under the Curve from Time Zero to Last Measurable Concentration (AUC0-t) of SEP-380135 and its Metabolites | Up to Day 11
Area Under the Curve from Time Zero to Infinity (AUCinfinity) of SEP-380135 and its Metabolites | Up to Day 11
Time to Maximum Concentration (Tmax) of SEP-380135 and its Metabolites | Up to Day 11

SECONDARY OUTCOMES:
Number of Participants With Treatment Emergent Adverse Events (TEAEs) | Up to 2 months
Number of Participants With Potentially Clinically Significant Changes in Vital Signs | Up to 2 months
Number of Participants With Potentially Clinically Significant Changes in Electrocardiogram (ECG) Parameters | Up to 2 months
Number of Participants With Potentially Clinically Significant Changes in Physical Examinations | Up to 2 months
Number of Participants With Potentially Clinically Significant Changes in Neurological Examinations | Up to 2 months
Number of Participants With Potentially Clinically Significant Changes in Clinical Laboratory Test Parameters | Up to 2 months
Number of Participants With Incidence of Suicidal Behavior, Suicidal Ideation and Suicidality Using the Columbia-Suicide Severity Rating Scale (C-SSRS) | Up to 2 months

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Vince Clinical Research, Overland Park, Kansas, United States

IPD SHARING:
Plan to Share IPD: No
Anonymized individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal. Small studies with less than 25 participants are excluded from data sharing.